CLINICAL TRIAL: NCT06894433
Title: Efficacy and Safety of NeuroEndoscopic Surgery for Large IntraCerebral Hemorrhage: a Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Efficacy and Safety of NeuroEndoscopic Surgery for Large IntraCerebral Hemorrhage
Acronym: NESICH 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Rong Hu, MD, Director of Department of Neurosurgery, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurosurg 05
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Intracerebral Haemorrhage
Keywords: intracerebral hemorrhage; neuroendoscopic; craniotomy
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Craniotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Neuroendoscopic Surgery to remove intracranial hematoma
  Interventions: Procedure: neuroendoscopic surgery
- Control Arm (Active Comparator): Craniotomy to remove intracranial hematoma
  Interventions: Procedure: craniotomy

INTERVENTIONS:
Procedure: neuroendoscopic surgery — Subjects will receive Neuroendoscopic Surgery followed by standard medical management
  Arms: Experimental Arm
Procedure: craniotomy — Subjects will receive Craniotomy followed by standard medical management
  Arms: Control Arm

SUMMARY:
This is a multicenter, randomized, controlled clinical trial comparing neuroendoscopic hematoma removal to craniotomy in the treatment of large intracerebral hemorrhage.

DETAILED DESCRIPTION:
Previous retrospective studies have demonstrated that neuroendoscopic surgery, compared to conventional craniotomy, significantly reduces operative duration and intraoperative blood loss, enhances hematoma evacuation rates, and improves postoperative outcomes, including neurological recovery, activities of daily living, and quality of life in patients with large cerebral hemorrhage. However, there is a paucity of prospective randomized controlled trials evaluating the efficacy of different surgical techniques for intracerebral hemorrhage. To address this gap, the investigators propose a multicenter, randomized, controlled clinical trial to compare the safety and efficacy of neuroendoscopic surgery versus craniotomy, aiming to provide evidence-based guidance for surgical decision-making in cerebral hemorrhage management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, male or female;
2. The time between onset and admission to the first diagnostic CT is within 24 hours (for no bystanders and the time of onset is unknown, the time of the last known patient in good condition is used);
3. Patients with supratentorial intracerebral hemorrhage (supratentorial intracerebral hemorrhage (supratentorial intracerebral hemorrhage) whose hematoma volume is ≥50ml or whose hematoma produces obvious space occupying effect and requires emergency surgery (including patients with cerebral hernia signs such as retarding or dilatation of light reflex of one pupil);
4. Before randomization, GCS score was 5-14, NIHSS score was ≥6;
5. mRS Before onset: 0-1 score;
6. Randomization within 24 hours after the first diagnostic CT;
7. The patient or family members are informed and voluntarily sign the informed consent;

Exclusion Criteria:

1. The clinical diagnosis is caused by cerebral aneurysm, cerebrovascular malformation, moyamoya disease, brain trauma, brain tumor, massive cerebral infarction hemorrhage transformation, coagulation dysfunction, etc.;
2. Thalamic hemorrhage, primary ventricular hemorrhage;
3. Platelet count <100×109/L, INR > 1.4;
4. Patients with advanced cerebral hernia (such as dilated bifidus and no light reflex) or unstable vital signs cannot tolerate surgery;
5. Irreversible brain stem impairment (eye fixation, bilateral pupil dilation), GCS≤4 points;
6. Any history of parenchyma or other intracranial subarachnoid, subdural or epidural blood and surgical history in the past 30 days;
7. Patients with severe advanced cognitive impairment (such as AD) or who are not expected to complete the follow-up plan as required;
8. Complicated with other serious diseases: including respiratory, circulation, digestion, urinary, endocrine, immune and blood systems;
9. Pregnant or breastfeeding women, or those who expect to become pregnant within one year;
10. are participating in other clinical trials (excluding: observational studies that do not involve intervention, natural history and/or epidemiological studies).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score 0-3 | 180 days
  Functional outcome (comparing the intervention group to the control), assessed with the modified Rankin Scale (mRS) at 6 months.The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) Score | 180 days
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
mortality | 30 days, 90 days and 180 days
  All cause mortality from onset to 180 days
Glasgow Outcome Scale Extended (GOS-E) | 180 days
  GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
Assessment of cognitive function with Mini-Mental State Examination (MMSE) | 90 days and 180 days
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function.
Quality of life measured with the 5-level EQ-5D (EQ-5D-5L) | 30 days and 180 days
  The EQ-5D-5L is a standard measure of health-related quality of life.EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state. The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health.
The proportion of patients with Modified Rankin Scale (mRS) score 0-2 | 180 days
  Functional outcome (comparing the intervention group to the control), assessed with the modified Rankin Scale (mRS) at 6 months.The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Length of ICU | Number of days from admission, up to 180 days
  Duration of stay in the ICU
Length of hospitalization | Number of days from admission to discharge, up to 180 days
  Duration of stay in the hospital
The proportion of patients with Modified Rankin Scale (mRS) score 0-3 | 30 days and 90 days
  Functional outcome (comparing the intervention group to the control), assessed with the modified Rankin Scale (mRS) at 6 months.The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Operation duration | From the beginning to the end of the surgery
  The length of the operation
Peroperative bleeding | During surgery
  The amount of blood lost during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rong Hu, MD, Study Chair — PLA Army Medical University
Locations (2):
- China (2):
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Dazhu County People's Hospital, Dazhou, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck J, Fung C, Strbian D, Butikofer L, Z'Graggen WJ, Lang MF, Beyeler S, Gralla J, Ringel F, Schaller K, Plesnila N, Arnold M, Hacke W, Juni P, Mendelow AD, Stapf C, Al-Shahi Salman R, Bressan J, Lerch S, Hakim A, Martinez-Majander N, Piippo-Karjalainen A, Vajkoczy P, Wolf S, Schubert GA, Hollig A, Veldeman M, Roelz R, Gruber A, Rauch P, Mielke D, Rohde V, Kerz T, Uhl E, Thanasi E, Huttner HB, Kallmunzer B, Jaap Kappelle L, Deinsberger W, Roth C, Lemmens R, Leppert J, Sanmillan JL, Coutinho JM, Hackenberg KAM, Reimann G, Mazighi M, Bassetti CLA, Mattle HP, Raabe A, Fischer U; SWITCH study investigators. Decompressive craniectomy plus best medical treatment versus best medical treatment alone for spontaneous severe deep supratentorial intracerebral haemorrhage: a randomised controlled clinical trial. Lancet. 2024 Jun 1;403(10442):2395-2404. doi: 10.1016/S0140-6736(24)00702-5. Epub 2024 May 15. PMID 38761811
- [Background] Pradilla G, Ratcliff JJ, Hall AJ, Saville BR, Allen JW, Paulon G, McGlothlin A, Lewis RJ, Fitzgerald M, Caveney AF, Li XT, Bain M, Gomes J, Jankowitz B, Zenonos G, Molyneaux BJ, Davies J, Siddiqui A, Chicoine MR, Keyrouz SG, Grossberg JA, Shah MV, Singh R, Bohnstedt BN, Frankel M, Wright DW, Barrow DL; ENRICH trial investigators; ENRICH Trial Investigators. Trial of Early Minimally Invasive Removal of Intracerebral Hemorrhage. N Engl J Med. 2024 Apr 11;390(14):1277-1289. doi: 10.1056/NEJMoa2308440. PMID 38598795
- [Background] Correction to: ICES (Intraoperative Stereotactic Computed Tomography-Guided Endoscopic Surgery) for Brain Hemorrhage: A Multicenter Randomized Controlled Trial. Stroke. 2017 Nov;48(11):e335. doi: 10.1161/STR.0000000000000153. No abstract available. PMID 29061841
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Background] Greenberg SM, Ziai WC, Cordonnier C, Dowlatshahi D, Francis B, Goldstein JN, Hemphill JC 3rd, Johnson R, Keigher KM, Mack WJ, Mocco J, Newton EJ, Ruff IM, Sansing LH, Schulman S, Selim MH, Sheth KN, Sprigg N, Sunnerhagen KS; American Heart Association/American Stroke Association. 2022 Guideline for the Management of Patients With Spontaneous Intracerebral Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2022 Jul;53(7):e282-e361. doi: 10.1161/STR.0000000000000407. Epub 2022 May 17. No abstract available. PMID 35579034
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Mendelow AD, Gregson BA, Fernandes HM, Murray GD, Teasdale GM, Hope DT, Karimi A, Shaw MD, Barer DH; STICH investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial intracerebral haematomas in the International Surgical Trial in Intracerebral Haemorrhage (STICH): a randomised trial. Lancet. 2005 Jan 29-Feb 4;365(9457):387-97. doi: 10.1016/S0140-6736(05)17826-X. PMID 15680453
- [Background] Teo KC, Fong SM, Leung WCY, Leung IYH, Wong YK, Choi OMY, Yam KK, Lo RCN, Cheung RTF, Ho SL, Tsang ACO, Leung GKK, Chan KH, Lau KK. Location-Specific Hematoma Volume Cutoff and Clinical Outcomes in Intracerebral Hemorrhage. Stroke. 2023 Jun;54(6):1548-1557. doi: 10.1161/STROKEAHA.122.041246. Epub 2023 May 22. PMID 37216445
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Huster G. Volume of intracerebral hemorrhage. A powerful and easy-to-use predictor of 30-day mortality. Stroke. 1993 Jul;24(7):987-93. doi: 10.1161/01.str.24.7.987. PMID 8322400
- [Background] Sondag L, Schreuder FHBM, Boogaarts HD, Rovers MM, Vandertop WP, Dammers R, Klijn CJM; Dutch ICH Surgery Trial Study Group, part of the CONTRAST consortiumdagger. Neurosurgical Intervention for Supratentorial Intracerebral Hemorrhage. Ann Neurol. 2020 Aug;88(2):239-250. doi: 10.1002/ana.25732. Epub 2020 Apr 30. PMID 32239722
- [Background] Ma L, Hu X, Song L, Chen X, Ouyang M, Billot L, Li Q, Malavera A, Li X, Munoz-Venturelli P, de Silva A, Thang NH, Wahab KW, Pandian JD, Wasay M, Pontes-Neto OM, Abanto C, Arauz A, Shi H, Tang G, Zhu S, She X, Liu L, Sakamoto Y, You S, Han Q, Crutzen B, Cheung E, Li Y, Wang X, Chen C, Liu F, Zhao Y, Li H, Liu Y, Jiang Y, Chen L, Wu B, Liu M, Xu J, You C, Anderson CS; INTERACT3 Investigators. The third Intensive Care Bundle with Blood Pressure Reduction in Acute Cerebral Haemorrhage Trial (INTERACT3): an international, stepped wedge cluster randomised controlled trial. Lancet. 2023 Jul 1;402(10395):27-40. doi: 10.1016/S0140-6736(23)00806-1. Epub 2023 May 25. PMID 37245517
- [Background] Pinho J, Costa AS, Araujo JM, Amorim JM, Ferreira C. Intracerebral hemorrhage outcome: A comprehensive update. J Neurol Sci. 2019 Mar 15;398:54-66. doi: 10.1016/j.jns.2019.01.013. Epub 2019 Jan 14. PMID 30682522
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944